CLINICAL TRIAL: NCT06367101
Title: Investigate the Effect of AR Environment Stimulation on Gait, Anxiety and Brain Connectivity of Individuals With Parkinson Disease
Brief Title: AR Stimulation Effects on Gait, Anxiety, and Brain Connectivity in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202002525B0
Record Dates: First submitted 2024-03-28; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease(PD)
Keywords: Augmented Reality; Heart rate variability; Gait; Stress
MeSH Terms: conditions — Parkinson Disease | interventions — Gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1:Healthy people (No Intervention): To establish baseline and reliability.
- Stage 2: PD people (No Intervention): To establish stage 3 training protocol.
- Stage 3: PD AR training group (Experimental): AR training with gait and HRV feedback
  Interventions: Other: AR training with gait and HRV feedback
- Stage 3: PD Control group (No Intervention): PD Control

INTERVENTIONS:
Other: AR training with gait and HRV feedback — Use projection-based AR system to train gait and HRV. To give gait and HRV feedback for subjects after AR training.
  Other Names: AR training group
  Arms: Stage 3: PD AR training group

SUMMARY:
A project aims at addressing gait impairments and non-motor symptoms such as anxiety and stress in Parkinson's disease (PD) patients through a novel approach involving heart rate variability (HRV) feedback and Augmented Reality (AR) training. The project is based on the premise that improving HRV, which reflects the adaptability of the autonomic nervous system, can enhance both motor functions like gait and non-motor symptoms.

DETAILED DESCRIPTION:
Gait impairments are prevalent among individuals diagnosed with Parkinson's disease (PD), presenting as shuffling steps, diminished stride length, increased cadence, freezing of gait, etc. Concurrently, non-motor symptoms, including anxiety, stress, and sleep disturbances, exert a substantial impact on the overall quality of life for PD patients.

Improving heart rate variability (HRV) can positively improve both motor and non-motor symptoms in PD. HRV serves as a reflective measure of the adaptability of the autonomic nervous system, a critical regulator of bodily functions, including gait. Diminished HRV correlates with impaired autonomic function, contributing to the observed gait abnormalities in individuals with Parkinson's disease. Training with HRV feedback has been shown to improve gait performance, stress, and anxiety.

The motor skill taxonomy proposed by Gentile seems to constitute just such a template for rehabilitation programs because it provides a two-dimensional basis for classifying a variety of motor skills. Meanwhile, AR offers a unique platform for creating intricate laboratory environments that facilitate non-invasive evaluation and rehabilitation, enabling the measurement of changes in the autonomic nervous system in response to environmental stimuli. Therefore, an Augmented Reality (AR) training program based on Gentile's theory, incorporating gait and HRV feedback and addressing PD-specific variables, will be developed.

The overarching goal of this 3-year project is to establish an effective environmental stimulation paradigm capable of ameliorating both motor and non-motor symptoms. This paradigm aims to contribute to the creation of tailored rehabilitation programs for individuals with Parkinson's disease. The project's progression is outlined as follows:

The first year: Design a standard AR environment based on Gentile's theory and establish test-retest reliability with 20 healthy subjects.

The second year: Test 30 individuals with PD in both real and AR environments to establish the relationship between different environmental stimuli for PD patients.

The third year: Randomize 30 individuals with PD into the AR training group and a control group. Evaluate the distinct training effects, with a focus on gait performance, gait initiation, freezing of gait, and anxiety levels.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

* Musculoskeletal injuries on legs.
* Osteoporosis.

PD subjects:

Inclusion Criteria:

- Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Walking Speed | Baseline and 6 weeks
  The time taken by participants to walk a standardized distance, typically expressed in centimeters per second (cm/s).
Step Length | Baseline and 6 weeks
  The linear distance between the two ankles, typically expressed in centimeter(cm).
Step Time | Baseline and 6 weeks
  The duration taken for one complete step, measuring from foot-off of one foot to the next foot-off of the same foot, usually expressed in seconds.
Time-Domain Index of Heart Rate Variability (HRV)：Standard deviation of RR intervals (SDRR) | Baseline and 6 weeks
  SDRR is the standard deviation of all recorded RR intervals (the time between successive heartbeats) over a specific period, usually expressed in milliseconds. This measure captures the total variability in heart rate, representing the physiological responses to a variety of internal and external stimuli. High SDRR values generally indicate greater heart rate variability, which is associated with good cardiovascular health and resilience to stress.
Time-Domain Index of HRV：pNN50 | Baseline and 6 weeks
  Percentage of successive RR intervals that differ by more than 50 ms. pNN50 reflects beat-to-beat variance in heart rate and is considered an indicator of parasympathetic nervous system activity, specifically linked to vagal tone. A higher pNN50 typically indicates better heart rate variability and healthier autonomic function.
Time-Domain Index of HRV：Root mean square of successive RR interval differences (RMSSD) | Baseline and 6 weeks
  RMSSD is the square root of the mean of the squares of successive differences between adjacent RR intervals. It emphasizes the high-frequency variations in heart rate that are typically mediated by the parasympathetic nervous system.
Frequency-Domain Index of HRV: Low Frequency (LF) | Baseline and 6 weeks
  The LF component typically represents the power of the HRV spectrum in the frequency range of 0.04 to 0.15 Hz. It is measured in milliseconds squared (ms²) or normalized units and is often interpreted as reflecting both sympathetic and parasympathetic activity,
Frequency-Domain Index of HRV: High Frequency (HF) | Baseline and 6 weeks
  HF typically covers the frequency range from 0.15 to 0.40 Hz and is associated with the respiratory cycle. HF power is usually measured in milliseconds squared (ms²) or normalized units and is indicative of the modulation of heart rate by the parasympathetic nervous system during breathing.
Frequency-Domain Index of HRV: Ratio of LF to HF Power | Baseline and 6 weeks
  The ratio of LF (low frequency) to HF power in the HRV spectrum. Since LF can represent both sympathetic and parasympathetic activity, comparing it to HF offers insights into the sympathetic-parasympathetic balance.
Total Time to Complete the Time Up and Go test (TUG test) | Baseline and 6 weeks
  The time, in seconds, it takes for a participant to complete the TUG test from the initial sitting position to returning to the seated position.

SECONDARY OUTCOMES:
Double Support Time | Baseline and 6 weeks
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Single Support Time | Baseline and 6 weeks
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle.
Swing Time | Baseline and 6 weeks
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds
Stance Time | Baseline and 6 weeks
  The portion of the gait cycle when the foot is in contact with the ground, supporting body weight. It's typically expressed as a percentage of the total gait cycle or in seconds
Cadence | Baseline and 6 weeks
  The number of steps an individual takes per minute, providing an overview of gait speed and rhythm, , expressed as steps per minute.
Total UPDRS-III Score | Baseline and 6 weeks
  The Unified Parkinson's Disease Rating Scale (UPDRS) Part III, also known as the UPDRS-III or the Motor Examination, is a critical component of the UPDRS used to assess the motor symptoms of Parkinson's disease (PD). To provide a comprehensive assessment of motor function in individuals with Parkinson's disease, covering aspects such as bradykinesia (slowness of movement), rigidity, tremors, and postural instability. The UPDRS-III consists of 14 items, each rated on a scale from 0 (normal) to 4 (severe), with a total possible score range from 0 to 108. Higher scores indicate greater motor impairment.
Total NFOG-Q Score | Baseline and 6 weeks
  The New Freezing of Gait Questionnaire (NFOG-Q) is a specialized tool designed to quantify the severity and impact of freezing of gait (FOG) episodes in individuals with Parkinson's disease (PD). To assess the presence, severity, and impact of FOG in individuals with Parkinson's disease, focusing on how it affects daily activities and mobility. The scores from Parts 2 and 3 are used to calculate a total score that reflects the overall severity and impact of FOG. This total score can help in gauging the effectiveness of treatments aimed at reducing the severity or frequency of FOG episodes.
Overall PDQ-39 Score | Baseline and 6 weeks
  To evaluate the quality of life across multiple dimensions affected by Parkinson's disease, including mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort. The PDQ-39 consists of 39 items, with each item relating to an aspect of life potentially impacted by PD. Responses to these items are aggregated into eight scales corresponding to the dimensions mentioned above.Each item is scored on a scale from 0 (never) to 4 (always), with the total score for each dimension being converted to a 0-100 scale. A higher score indicates a lower quality of life.
Total HADS Score | Time Frame: Baseline and 6 weeks.
  The Hospital Anxiety and Depression Scale (HADS) is a validated instrument designed to identify and quantify the severity of anxiety and depression symptoms, particularly focusing on the psychological rather than the somatic aspects to avoid confounding with physical illnesses. To screen for, and evaluate the severity of, anxiety and depression symptoms in a wide range of healthcare settings, especially useful in populations where physical illness might overlap with psychological distress. The scores for each subscale (anxiety and depression) range from 0 to 21. These can be combined to give a total HADS score, which ranges from 0 to 42, with higher scores indicating more severe symptoms.
Overall PSQI Score | Time Frame: Baseline and 6 weeks.
  The Pittsburgh Sleep Quality Index (PSQI) is a comprehensive self-rated questionnaire that assesses sleep quality and disturbances over the past month. To evaluate the quality and patterns of sleep, identifying sleep disorders and quantifying the degree of sleep-related problems. Each component is scored on a scale of 0 to 3, with the total PSQI score ranging from 0 to 21. Higher scores indicate poorer sleep quality.
Non-linear Index of HRV: SD1 | Baseline and 6 weeks
  SD1 is calculated from the Poincaré plot, where it measures the dispersion of points perpendicular to the line of identity, usually expressed in milliseconds. This dispersion specifically quantifies the short-term variability in heart rate, primarily influenced by the parasympathetic nervous system. SD1 provides insight into the rapid changes in heart rate variability, offering a unique perspective on autonomic nervous system activity that traditional time-domain and frequency-domain measures might not fully capture.
Non-linear Index of HRV: SD2 | Baseline and 6 weeks
  SD2 is calculated as the standard deviation of points along the line of identity in the Poincaré plot, reflecting long-term heart rate variability, usually expressed in milliseconds. This measure captures broader fluctuations in heart rate that are influenced by both sympathetic and parasympathetic nervous system activities. SD2 provides insights into the overall autonomic balance and the body's ability to adapt to sustained physiological stressors or environmental changes. It is particularly useful in studies investigating chronic stress, cardiovascular health, or the impact of long-term interventions.
Non-linear Index of HRV: Ratio of SD1-to-SD2 | Baseline and 6 weeks
  The SD1/SD2 ratio is calculated by dividing SD1, which measures short-term variability and is predominantly influenced by parasympathetic activity, by SD2, which measures long-term variability and reflects both sympathetic and parasympathetic influences. This ratio is useful for assessing the autonomic balance or the sympathetic-parasympathetic interaction. A higher SD1/SD2 ratio indicates a dominance of parasympathetic activity relative to sympathetic, suggesting a more "relaxed" autonomic state, whereas a lower ratio indicates a relative dominance of sympathetic activity, which could be associated with stress, reduced cardiac health, or other health risks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No